CLINICAL TRIAL: NCT03438838
Title: Randomised Clinical Trial Comparing Relief of Dysphagia Between Laparoscopic Heller's Myotomy Alone Versus Laparoscopic Heller's Myotomy With Anterior Fundoplication In Achalasia Cardia-A Pilot Study
Brief Title: Randomised Trial Between LHM Alone Vs LHM With Anterior Fundoplication In Achalasia Cardia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Principal Investigator, Hirdaya H Nag, MS, Dr. Prof, Govind Ballabh Pant Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIPMER
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Achalasia Cardia
Keywords: Achalasia, LHM, Anterior fundoplication
MeSH Terms: conditions — Esophageal Achalasia | interventions — Heller Myotomy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be randomized using computer generated table of random numbers contained in a sealed opaque envelope to be opened in operation theatre after induction anesthesia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Heller's Myotomy (LHM)alone (Active Comparator): A minimum 10 patients undergo Laparoscopic Heller's myotomy alone
  Interventions: Procedure: Laparoscopic Heller's myotomy
- LHM with Anterior Fundoplication (Active Comparator): A Minimum 10 patients undergo Laparoscopic Heller's myotomy along with fundoplication
  Interventions: Procedure: Laparoscopic Heller's myotomy; Procedure: Anterior Fundoplication

INTERVENTIONS:
Procedure: Laparoscopic Heller's myotomy — Laparoscopic Heller's myotomy:
  Anterior wall of esophagus is exposed by opening peritoneum and minimal dissection of fat over it. Myotomy is started at 2 cm above the esophago- gastric junction. Initial plane is created using dissector and further muscles are split using pair of dissector or bowel holding forceps for length of 7 to 8 cm with 2 cm over stomach
Procedure: Anterior Fundoplication — The Fundus was sutured with 3 stitches on either side of the esophagus to right and left crus of diaphragm using ethibond(1-0) beside intervening stitch over esophagus. Width of fundoplication is kept approximately at 2cm. The proximal short gastric vessels were divided only if the fundus is insufficiently mobile
  Arms: LHM with Anterior Fundoplication

SUMMARY:
Back ground: Achalasia Cardia (AC) manifests with major symptom dysphagia. Surgery as the treatment modality relieves dysphagia in most of the patients. Laparoscopic Heller's myotomy(LHM) is the surgery of choice but is associated with gastroesophageal reflux. Anterior fundoplication (Dor Fundoplication) is usually combined with LHM in patients with AC. It reduces gastroesophageal reflux following LHM. It has been observed that along with reduction of gastroesophageal reflux Dor Fundoplication also affects relief of dysphagia. But it has not been prospectively studied.

Hypothesis:The hypothesis of present study is that "Frequency of dysphagia following Laparoscopic Heller's myotomy with Dor fundoplication is more than that compared to Laparoscopic Heller's myotomy alone in patients with Achalasia Cardia".

Methods: From December2017 to November 2018 minimum of 20 patients with diagnosis of Achalasia cardia will be randomized to receive either Laparoscopic Heller's myotomy (LHM) alone or LHM with Dor fundoplication. Symptomatic outcomes would be assessed using frequency of dysphagia and Eckardt's score. .

Outcomes: Primary outcome is Frequency of dysphagia and secondary outcome is manometry pressure assessment. Statistical analysis would be done using Statistical Package for the Social Sciences (SPSS) soft ware. P value < 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 years or more) with Achalasia cardia

Exclusion Criteria:

* Patients of achalasia with axis deviation
* Patients with history of pneumatic dilatation
* Patient with other associated motility or non motility disorders
* Patients with pseudoachalasia Prior gastric or esophageal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Dysphagia | Minimum one month after surgery
  None- 0 Occasional-1 Daily-2 Each meal-3

SECONDARY OUTCOMES:
Manometry pressure | Minimum one month after surgery
  Using High resolution Manometry
Gastro esophageal reflux | Minimum after one month
  GERD symptoms
Eckardt's score | Minimum after one month
  Dysphagia
  * 0-None
  * 1-Occasional
  * 2-Daily
  * 3-Each meal Retrosternal pain
  * 0-None
  * 1-Occasional
  * 2-Daily
  * 3-Each meal Regurgitation
  * 0-None
  * 1-Occasional
  * 2-Daily
  * 3-Each meal Weight loss
  * 0-None
  * 1-less than 5 kg
  * 2-5 to 10kg
  * 3-more than 10kg
  Minimum score: 0 Maximum score: 12

CONTACTS AND LOCATIONS:
Overall Officials: Hirdaya H Nag, MS, Principal Investigator — GIPMER
Locations (1):
- GIPMER, New Delhi, India

IPD SHARING:
Plan to Share IPD: No